CLINICAL TRIAL: NCT01770184
Title: Clinical Effectiveness of Self-Management Education Post-Mild Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1K23HD073190-01 (NIH)
Record Dates: First submitted 2013-01-11; First posted 2013-01-17 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Stroke; Chronic Disease
Keywords: Self-management; Rehabilitation; Occupational Therapy
MeSH Terms: conditions — Stroke; Chronic Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will receive the rehabilitation services and support that is recommended and provided in the current health care structure. The intervention group will also receive the Chronic Disease Self-Management Program (CDSMP). The CDSMP is an education program based on the concept of self-management. Self-management refers to the ability of an individual to manage the day-to-day responsibilities of living with a chronic condition. The CDSMP will be delivered in two and a half hour sessions, once a week, for six weeks, in group format.
  Interventions: Behavioral: Chronic Disease Self-Management Program (CDSMP)
- Usual Care Group (No Intervention): The usual care group for this study will receive the rehabilitation services and support that is recommended and provided in the current health care structure. No additional intervention will be provided to the usual care group within this study.

INTERVENTIONS:
Behavioral: Chronic Disease Self-Management Program (CDSMP)
  Arms: Intervention Group

SUMMARY:
Individuals who have a mild stroke have a 44% risk of dying from a second stroke within 10 years which is in large part due to the cyclical relationship of chronic disease, poor health, and mild stroke which has gone largely unnoticed in the United States. Self-management intervention has been proven to be an effective intervention to increase healthy behaviors, improve overall health status, decrease healthcare utilization/cost, decrease depressive symptoms, and improve participation in people with a variety of chronic conditions; however, it has never be used with individuals with mild stroke. The critical next step and goal of this study is to evaluate if self-management intervention will improve health outcomes for persons with mild stroke. The overall hypothesis of this study is that self-management intervention will improve outcomes in the mild-stroke population.

ELIGIBILITY:
Inclusion Criteria:

* a mild stroke as NIHSS total scores 0-5
* 18-90 years of age
* English speaking
* identified as having at least one other chronic condition besides stroke

Exclusion Criteria:

* severe aphasia (NIHSS aphasia score=2)
* moderate to severe cognitive impairment (MOCA < 21)
* history of dementia
* hemorrhagic stroke
* neurological diagnoses other than stroke
* major psychiatric illness (A diagnosis of bipolar disorder, obsessive compulsive disorder, panic disorder, schizophrenia, post-traumatic stress disorder, and borderline personality disorder)
* a score of no-higher than 20 on the PHQ-9 indicating significant depressive symptoms
* terminal illness

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Adapted Illness Intrusiveness Ratings (AIIR) | Change from baseline to 6-months post-stroke
Healthcare Utilization Survey (HCUS) | Change from baseline to 6-months post-stroke

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Change from baseline to 6-months post-stroke
Work Ability Index (WAI) | Change from baseline to 6-months post-stroke
Reintegration to Normal Living Index (RNLI) | Change from baseline to 6-months post-stroke
World Health Organization Quality of Life (WHOQOL-BREF) | Change from baseline to 6-months post-stroke
Chronic Disease Self-Efficacy Scale (CDSES) | Change from baseline to 6-months post-stroke
Multidimensional Assessment of Fatigue (MAF) | Change from baseline to 6-months post-stroke
Activity Card Sort (ACS) | Change from baseline to 6-months post-stroke
Stroke Impact Scale (SIS) | Change from baseline to 6-months post-stroke

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Wolf, OTD, MSCI, OTR/L, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, School of Medicine, Program in Occupational Therapy, St Louis, Missouri, United States

REFERENCES:
- [Derived] Crocker TF, Brown L, Lam N, Wray F, Knapp P, Forster A. Information provision for stroke survivors and their carers. Cochrane Database Syst Rev. 2021 Nov 23;11(11):CD001919. doi: 10.1002/14651858.CD001919.pub4. PMID 34813082
- See also: Performance, Participation, and Neurorehabilitation Laboratory: Timothy J. Wolf, OTD, MSCI, OTR/L (PI) — http://ot.wustl.edu/ot/otweb.nsf/6c18fc53358d390286256cde00604464/7f1c60fc33a21e2686257a8b0056d6f5?OpenDocument